CLINICAL TRIAL: NCT01942772
Title: Design of A Powered Ankle Foot Orthoses for Ankle Rehabilitation
Brief Title: A Powered Ankle Foot Rehabilitation Orthosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Beijing Institute of Technology (Other)
Collaborators: China Rehabilitation Research Center (Other Government)
Responsible Party: Principal Investigator, Yang Bai, researcher, Beijing Institute of Technology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: byang421
Record Dates: First submitted 2013-08-27; First posted 2013-09-16 (Estimated); Last update posted 2013-09-16 (Estimated); Status verified 2013-03

CONDITIONS: Stroke; Ankle Injuries
Keywords: powered ankle-foot orthosis; mechanical structure; optimization; dorsiflexion; plantar flexion; gait; servomotor; ankle rehabilitation
MeSH Terms: conditions — Stroke; Ankle Injuries

ARMS (1):
- experimental test of healthy subjects (Experimental): wearing experiment，motion experiment
  Interventions: Device: Ankle-Foot Orthosis

INTERVENTIONS:
Device: Ankle-Foot Orthosis

SUMMARY:
Ankle rehabilitation training becomes a tough question for the patients with ankle joint injuries especially with the hemiplegia after stroke. Here a novel powered ankle foot orthoses which can provide ankle dorsiflexion and plantar flexion assistant using electric motor is proposed in this paper. The mechanical structure of the orthoses includes wearing parts, ankle joint hinged part, driving unit, transmission mechanism and sensing units. This study provides a new method for ankle foot orthoses design and has great significance for ankle rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* ankle joint injuries about dorsiflexion and plantar flexion
* Ability to keep balance independently

Exclusion Criteria:

* ankle joint injuries about varus and valgus rehabilitation
* two assistants needed while walking

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2 (Estimated)
Dates: Start 2013-01; Primary Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
good performance of the ankle foot orthosis | one month
  Two researchers wore the ankle foot orthosis without any motion to test the rationality of design size and wearing coordination；motion experiment without load was carried out to test the stability of transmission structure and effectiveness of motor control. The ankle foot orthosis was fixed on a table.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Institute of Technology, Beijing, Beijing Municipality, China

REFERENCES:
- See also: WalkAide Compared to Ankle-Foot Orthosis (AFO) in Stroke Patients — http://clinicaltrials.gov/ct2/show/NCT01087957?term=ankle-foot+orthosis&rank=1
- See also: Rehabilitation of Early Stroke Patients Using an AFO: an RCT — http://clinicaltrials.gov/ct2/show/NCT01006772?term=ankle-foot+orthosis&rank=3